CLINICAL TRIAL: NCT05665478
Title: Dose Optimization of Carbapenem Antibacterials in Febrile Neutropenia Patients Based on PPK/PD Model and MAPB Method and Research on Individualized Drug Use Software
Brief Title: Population Pharmacokinetics/Pharmacodynamics of Carbapenems in Febrile Neutropenia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-LCYJ-PY-48
Record Dates: First submitted 2022-11-20; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-11

CONDITIONS: Febrile Neutropenia; Pharmacokinetics; Pharmacodynamic; Carbapenems
MeSH Terms: conditions — Febrile Neutropenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- model intervention group (Active Comparator): The model was used for prediction to guide the later dosing regimen
  Interventions: Other: Dose prediction using population pharmacokinetic models
- Non-intervention group (No Intervention): In the non-intervention group, the doctor chose the treatment plan.

INTERVENTIONS:
Other: Dose prediction using population pharmacokinetic models — Dose prediction using population pharmacokinetic models.
  Arms: model intervention group

SUMMARY:
1. Evaluating the differences in the efficacy and safety of meropenem optimal dosing regimen predicted by the PPK/PD model combined with MAPB method for patients with malignant hematological myelopathy accompanied by fever, as compared with the current conventional treatment regimen;
2. The visualization software of meropenem individualized medication was developed with the help of JAVA development language, J2EE framework and SQL Server database.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, regardless of gender;
2. Patients with malignant hematological diseases with neutropenia and fever are judged as high-risk patients according to the Guidelines for Clinical Application of Antibiotics in Patients with Neutropenia and Fever in China (2020 Edition);
3. There is infection, and the results of drug sensitivity test show that pathogenic bacteria are sensitive to meropenem or meropenem is used according to experience;
4. The blood concentration of meropenem has reached a steady state;
5. Each patient's blood sample points ≥2, and cases with only one blood sample point can also be included in the database;
6. Sign the informed consent form.

Exclusion Criteria:

1. Patients with non-malignant hematological diseases;
2. Non-granular deficiency with fever;
3. Those who did not reach steady state when receiving meropenem;
4. There is a history of meropenem drug allergy;
5. The patient lacks treatment compliance based on the patient's history and the judgment of the researcher;
6. The patient has hemophagocytic syndrome;
7. Patients undergoing renal replacement therapy;
8. Patients with incomplete clinical evaluation data (such as lack of information on renal function and biochemical indicators, and inability to obtain blood samples);
9. The sample contains components that interfere with the determination of drug concentration (such as valproic acid and chloramphenicol);
10. Pregnant and lactating women;
11. Cases considered by the researcher as unsuitable for inclusion.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of antipyretic time 12 days after drug administration | Baseline and at the first 0 hour, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours, 144 hours, 168 hours, 192 hours, 216 hours, 240 hours, 264 hours, 288 hours after administration,
  The antipyretic time of the experimental group is compared with that of the control group. If the antipyretic time of the experimental group is shorter than that of the control group, the experimental treatment is considered effective.

CONTACTS AND LOCATIONS:
Overall Officials: Yudong Qiu, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School